CLINICAL TRIAL: NCT06752135
Title: Node Positive Cervical Cancer Treated by Neoadjuvant Chemotherapy Plus Radical Surgery: a Single Center Experience
Acronym: HRCC1
Status: Terminated | Type: Observational
Why Stopped: Retrospectively data collection complited
Sponsor: Azienda Policlinico Umberto I (Other)
Collaborators: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Innocenza Palaia, Professor, Azienda Policlinico Umberto I
Other Study IDs: AOU Umberto I; Cx - Prot.0330/2024|Rif. 7350 (Other: Azienda Policlinico Umberto I)
Record Dates: First submitted 2024-12-09; First posted 2024-12-30 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Cervical Carcinoma
Keywords: cervical carcinoma; neoadjuvant chemotherapy.; observational study; retrospective; radiological prognostic factors; imaging methodologies; MRI; TC scan; PFS; OS; pathological parameters; radiological parameters; clinical parameters
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Conization; Magnetic Resonance Imaging; Neoadjuvant Therapy; Cisplatin; Carboplatin; Paclitaxel; Hysterectomy; Salpingo-oophorectomy; Lymph Node Excision; Brachytherapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cervical squamous cell carcinoma or adenocarcinoma (FIGO IIIC1-2): The study cohort included women aged 18-75 years with histologically confirmed cervical squamous cell carcinoma or adenocarcinoma, positive lymph nodes (FIGO IIIC1-2), no prior oncological treatments, no pregnancy, a performance status of 0-2 (WHO), life expectancy of at least 3 months, and no evidence of distant metastasis or concomitant cancers.
  Interventions: Procedure: cervical biopsies/conization,; Diagnostic Test: imaging tests (TCTB, TC-PET, MRI); Drug: neoadjuvant chemotherapy (cisplatin or carboplatin plus paclitaxel); Procedure: hysterectomy, salpingo-oophorectomy, and lymphadenectomy; Radiation: brachytherapy

INTERVENTIONS:
Procedure: cervical biopsies/conization, — Diagnostic laparoscopy was used in selected cases to evaluate potential peritoneal spread.
Diagnostic Test: imaging tests (TCTB, TC-PET, MRI) — The staging procedures included imaging such as chest CT, abdomino-pelvic MRI, and PET-CT to assess tumor spread and lymph node involvement.
Drug: neoadjuvant chemotherapy (cisplatin or carboplatin plus paclitaxel) — Patients received three cycles of platinum-based neoadjuvant chemotherapy (cisplatin or carboplatin plus paclitaxel), followed by imaging to assess treatment response.
Procedure: hysterectomy, salpingo-oophorectomy, and lymphadenectomy — Eligible patients underwent radical surgery, including hysterectomy, salpingo-oophorectomy, and lymphadenectomy, with adjuvant therapy administered as needed based on surgical findings. Follow-up included regular clinical exams, imaging, and tests to monitor for recurrence.
Radiation: brachytherapy — alternative to cCRT-B.

SUMMARY:
This clinical study focuses on the treatment of high-risk locally advanced cervical cancer (LACC) in women with lymph node involvement (stages IIIC1 and IIIC2). Cervical cancer (CC) is a significant health concern worldwide, particularly for women, with high rates of diagnosis and mortality. While there have been advances in prevention and treatment, a substantial number of patients are still diagnosed with advanced-stage disease, which often involves cancer spread to nearby lymph nodes.

In standard practice, patients with LACC are usually treated with chemoradiation plus brachytherapy (cCRT-B). However, this approach can have considerable side effects and doesn't always provide a long-term cure. The study explores an alternative treatment regimen involving neoadjuvant chemotherapy (NACT) followed by radical surgery (RS) to evaluate its potential in improving survival outcomes and reducing recurrence. Neoadjuvant chemotherapy, a treatment given before surgery to shrink tumors, is often used for different types of cancer, and this study examines its benefits in cervical cancer patients with nodal involvement.

The main goal of this study is to determine whether NACT combined with radical surgery can offer survival rates and progression-free survival comparable to the standard treatment of chemoradiation. Additionally, the study aims to assess patterns of recurrence after treatment and to explore how these patients responded to further treatment options.

Study hypotheses: NACT + RS as a viable alternative: The hypothesis is that the combination of NACT followed by radical surgery may lead to survival outcomes comparable to those achieved by the standard cCRT-B treatment, particularly in patients with node-positive cervical cancer.

Improved recurrence management: Another key hypothesis is that the recurrence patterns in patients treated with NACT + RS are different, and a significant proportion of recurrent cases may be treated successfully with curative approaches such as surgery or radiotherapy.

Quality of life considerations: This treatment approach may offer better quality of life compared to chemoradiation by avoiding some of the severe side effects of radiotherapy, such as vaginal stenosis and other complications.

The study follows 97 patients who were treated at the Gynecologic Oncology Unit of Policlinico Umberto I, Sapienza University of Rome, between 2012 and 2022. The patients were diagnosed with cervical cancer and were in stages IIIC1 or IIIC2, meaning they had lymph node involvement. These patients received three cycles of chemotherapy (cisplatin and paclitaxel) followed by radical surgery, with further treatment depending on the surgical outcomes. After surgery, patients underwent a follow-up program to monitor for disease recurrence and overall survival.

DETAILED DESCRIPTION:
This study is a retrospective observational investigation aimed at evaluating the treatment outcomes of neoadjuvant chemotherapy (NACT) followed by radical surgery (RS) in patients with high-risk locally advanced cervical cancer (LACC) exhibiting positive lymph nodes (FIGO IIIC1-2 stage). The study analyzes recurrence patterns, subsequent treatments, and survival outcomes in a cohort of patients treated over a 10-year period at the Gynecologic Oncology Unit of Policlinico Umberto I, Sapienza University of Rome.

Study objectives and hypotheses: the primary hypothesis of this study is that the combination of NACT and radical surgery can offer survival outcomes and patterns of recurrence comparable to the standard chemoradiotherapy (cCRT-B) for LACC patients with nodal involvement (FIGO IIIC1-2). The secondary hypothesis suggests that a significant proportion of patients with recurrent disease can benefit from curative interventions (surgery, chemotherapy, or chemoradiotherapy), improving overall survival (OS) and progression-free survival (PFS) rates.

Study design and methodology: this study involved 97 patients diagnosed with locally advanced cervical cancer, all treated with NACT followed by RS from January 2012 to December 2022. The study's inclusion criteria were: patients aged 18-75 years with histologically confirmed cervical squamous cell carcinoma or adenocarcinoma, positive lymph nodes (FIGO IIIC1-2), and no prior oncological treatments. The treatment protocol involved three cycles of platinum-based NACT (cisplatin or carboplatin plus paclitaxel), followed by imaging assessments to evaluate the response to chemotherapy. Only patients with complete or partial responses according to RECIST criteria were considered for subsequent radical surgery.

The study also assessed the pattern of recurrence, treatments for recurrence, and survival outcomes, with data collection including clinical examination, imaging (CT, MRI, PET-CT), and histopathological analyses. The main measures of success were OS and PFS, with statistical analyses conducted using Kaplan-Meier methods.

Quality assurance and data management: the study adhered to a rigorous quality assurance plan that ensured accurate data collection, validation, and analysis. Data were sourced from an institutional database and reviewed by an expert panel. To ensure consistency, data were cross-verified with external sources such as medical records, and discrepancies were resolved through audit procedures. A detailed data dictionary was maintained to ensure consistency in variable definitions, coding (e.g., WHO drug dictionary), and reporting standards.

Atatistical analysis: the statistical analysis involved the Fisher exact test for categorical data, t-tests for parametric continuous variables, and the Mann-Whitney U test for non-parametric data. Survival data were analyzed using the Kaplan-Meier method, estimating OS and PFS for all patients and subgroups, including comparisons based on FIGO stage IIIC1 versus IIIC2. Survival outcomes were also analyzed in relation to the recurrence sites (e.g., pelvic nodes, central pelvis).

ELIGIBILITY:
Inclusion Criteria:

* Women aged ≥ 18 years attending the AOU Policlinico Umberto I
* histological diagnosis of cervical squamous cell carcinoma or adenocarcinoma; presence of positive lymph nodes at imaging (FIGO IIIC1-2 stage);
* ECOG performance status 0 or 1;
* No previous oncological treatments;
* No actual pregnancy;
* Life expectancy of at least 3 months;
* Ability to understand and willingness of the subject to participate in the trial confirmed by the signature of the written informed consent.
* No of distant metastasis or concomitant neoplasms.

Exclusion Criteria:

* Patients who have a clinical diagnosis different from advanced cervical cancer stages IB2-IVA
* Patients who have not received neoadjuvant chemotherapy
* Systemic diseases or immunodeficiencies
* Patients who are HCV+, HBV+, or HIV+

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population consisted of women aged 18 years or older who attended the AOU Policlinico Umberto I and had been diagnosed with cervical cancer, specifically squamous cell carcinoma or adenocarcinoma. These women had imaging-confirmed positive lymph nodes, corresponding to FIGO stages IIIC1-2, indicating locally advanced disease. The patients were required to have an ECOG performance status 0-1, suggesting that they were in relatively good general health and able to tolerate treatment. Participants had no prior history of oncological treatments and were not pregnant at the time of enrollment. Eligible participants were expected to have a life expectancy of at least three months. Additionally, they needed to be capable of understanding the study and willing to provide written informed consent. Patients with distant metastases or other concomitant malignancies were excluded, as were those with conditions that could complicate treatment, such as systemic diseases, immunodeficiencies.
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2024-04-10 (Actual); Primary Completion 2024-08-08 (Actual); Study Completion 2024-12-06 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) in Patients with Cervical Cancer After NACT + Radical Surgery | Progression-Free Survival (PFS) were assessed at 2 years and 5 years after the treatment completion, with follow-up assessments conducted regularly every 3 months for the first 2 years and then every 6 months until the 5th years
  Progression-Free Survival (PFS) was measured as the proportion of patients surviving without death from any cause. Progression-Free Survival (PFS) was measured as the proportion of patients without disease progression after the treatment. Metrics were calculated for the entire cohort and by FIGO stage (IIIC1 and IIIC2). The survival analysis was performed using Kaplan-Meier estimation, and survival curves were presented for PFS. These outcomes were analyzed to assess the long-term effectiveness of NACT followed by radical surgery in cervical cancer patients.
Overall Survival (OS) in Patients with Cervical Cancer After NACT + Radical Surgery | Overall Survival (OS) were assessed at 2 years and 5 years after the treatment completion, with follow-up assessments conducted regularly every 3 months for the first 2 years and then every 6 months until the 5th years
  Overall Survival (OS) was measured as the proportion of patients surviving. Metrics were calculated for the entire cohort and by FIGO stage (IIIC1 and IIIC2). The survival analysis was performed using Kaplan-Meier estimation, and survival curves were presented for OS. These outcomes were analyzed to assess the long-term effectiveness of NACT followed by radical surgery in cervical cancer patients.

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Policlinico Umberto I - Roma, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided